CLINICAL TRIAL: NCT01035996
Title: Dopamine Function and Reward Processing In Schizophrenia
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905401; 05-DA-N401
Record Dates: First submitted 2009-12-18; First posted 2009-12-21 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2017-02-13

CONDITIONS: Schizophrenia
Keywords: Classical Conditioning; fMRI; Schizophrenia; TD Model; Incentive Salience
MeSH Terms: conditions — Schizophrenia

SUMMARY:
Background:

- Schizophrenia is associated with cognitive impairment in different parts of the brain, including those associated with learning and memory. The brain activity associated with these impairments, however, is poorly understood. Researchers are interested in studying how the brain chemical dopamine, which is involved in responding to incentives and rewards like money or food, works differently in the brains of people who have schizophrenia.

Objectives:

- To study reward processing in individuals with schizophrenia who are taking different types of medication, compared with healthy volunteers.

Eligibility:

- Individuals between 18 and 55 years of age who (a) have been diagnosed with schizophrenia/schizoaffective disorder and are taking the antipsychotic medication clozapine, (b), have been diagnosed with schizophrenia/schizoaffective disorder and are taking a different second-generation antipsychotic, or (c) are healthy volunteers.

Design:

* This study will involve one screening visit and one or more visits for testing and functional magnetic resonance imaging (fMRI) scans. During the screening visit, participants will complete questionnaires and provide information about their physical and psychological health.
* Participants will receive training in the tasks to be performed at the scanning sessions during the screening visit.
* During the fMRI scans, participants will complete one or two of four possible reward-based tasks:
* A task that enables participants to win money based on their response to a target item.
* A task that provides small amounts of juice over specific time intervals, followed by a procedure to be completed outside the scanner.
* A task that involves choosing figures or shapes and winning money based on responses.
* A game of chance involving predictions based on shapes shown on a screen.
* Participants will also provide blood samples for research and testing.

DETAILED DESCRIPTION:
Objective:

Schizophrenia (SC) is associated with cognitive impairment in a variety of domains, including learning and memory. The neural underpinnings of these cognitive deficits, however, are poorly understood. Based on evidence that abnormal functioning of brain dopamine (DA) systems is implicated in both schizophrenia and mechanisms of reinforcement processing, we proposed to test theories of the functional role of dopamine in schizophrenia. Specifically, the studies described here test two main ideas about DA function and its possible contribution to SC: 1) its role in facilitating learning of cue-reward associations; and 2) its role in signaling mismatches between expected and experienced outcomes (called prediction errors).

Study Population:

In order to assess brain responses to outcomes, and cues predictive of outcomes, we will enroll 135 total participants (SC patients and controls), aged 18 - 55. For a first set of experiments, we enrolled 54 total subjects (37 SCs and 17 controls) to achieve 34 total completers (24 SCs and 10 controls). In a second set of experiments, our goal is to examine two types of SC patients (those taking clozapine and those taking a different second-generation antipsychotic). For these experiments, we will enroll 81 total subjects (27 controls, 27 SCs taking clozapine, and 27 SCs taking a different second-generation antipsychotic) to achieve approximately 47 total completers (15 controls, 16 SCs taking clozapine, and 16 SCs taking a different second-generation antipsychotic).

Design:

We will measure brain activity using functional magnetic resonance imaging (fMRI), in conjunction with the performance of reinforcement processing tasks from the literature. These paradigms involve either the passive observation of reinforcement contingencies, or the requirement to make an appropriate response within a time window in order to earn positive feedback. The ongoing study uses two specific paradigms: one examining the impact of brain responses to feedback on subsequent learning, and one investigating how brain responses to a monetary reinforcer are modulated by the unexpectedness of the event.

Outcome Measures:

In the current study, we will investigate differences in MRI responses to outcomes between SC patients and controls, and between subgroups of patients. In particular, we are interested in determining whether MRI responses in components of reward circuits, such as the midbrain, basal ganglia, and orbitofrontal cortex, are attenuated in SC patients, in the context of paradigms that require individuals to detect mismatches between expected and experienced outcomes, and to modify responses based on those mismatches. We hypothesize that learning deficits in SC stem primarily from impairments in the signaling of errors in reward prediction, and that abnormalities in the signaling of errors in reward prediction will be reflected in abnormal stimulus-evoked activation in the primarily in two brain areas in SC patients (both DA target areas): prefrontal cortex and the neostriatum. We predict that these signals will relate systematically to performance on a reinforcement-learning task.

ELIGIBILITY:
* INCLUSION CRITERIA::

Individuals will be eligible for participation in one of the proposed experimental groups on the condition that they are:

1. Aged between 18 55 years.
2. In good health, based on history and physical examination
3. Right-handed (i.e. as assessed using the Edinburgh Handedness Inventory)

In addition, patient participants:

1. Must meet DSM-IV criteria for schizophrenia or schizoaffective disorder at the time of assessment, and
2. Must have had 4 weeks of stable pharmacological treatment (same medications at same doses).

Behavioral Subject Only:

1. Aged between 18 55 years.
2. In good health, based on history and physical examination
3. Right-handed (i.e. as assessed using the Edinburgh Handedness Inventory)

In addition, patient participants:

1. Must meet DSM-IV criteria for schizophrenia or schizoaffective disorder at the time of assessment, and
2. Must have had 4 weeks of stable pharmacological treatment (same medications at same doses).

Individuals will be eligible for participation in one of the proposed experimental groups on the condition that they are:

EXCLUSION CRIERIA:

Participants in MRI scanning experiements

All participants in the MRI scanning experiements will undergo standard screening as in the clinical policies of the IRP:

All Participants in the MRI scanning experiments

Participants in both experimental groups will be excluded from participation if they:

1. Are unable to undergo MRI scanning due to pregnancy (via pregnancy test), implanted or attached metallic devices (e.g. cardiac pacemaker or neurostimulator; some artificial joints metal pins; surgical clips; braces; or other implanted metal parts), claustrophobia, or syncope, by self-report;
2. Show current evidence of severe hypertension, as indicated by a blood pressure measurement at or above 190 systolic or 110 diastolic on two separate occasions. Potential participants with evidence of chronic and/or poorly controlled hypertension may be excluded by the MRP even with measurements below those values;
3. Show current evidence of diabetes, as indicated by a blood sugar measurement of over 300 mg/dl. Potential participants with evidence of chronic and/or poorly controlled diabetes may be excluded by the MRP even with measurements below those values;
4. Suffer from HIV infection, coagulopathies, or other major medical illness which, in the judgment of the MRP, would seriously compromise the quality of the data gathered;
5. Have any neurological illnesses that would interfere with the quality of the neuroimaging data gathered, i.e. to include (but not limited to): seizure disorders; migraine; multiple sclerosis; movement disorders; or history of head trauma, CVA, or CNS tumor;
6. Are notably cognitively impaired by history or observation;
7. Have a DSM-IV diagnosis of past alcohol or substance dependence (with the exception of nicotine);
8. Test positively for any of 7 common banned substances at the time of screening;
9. Are lactating, as hormonal fluctuations associated with lactation may interact with dopamine system function.

Normal, Healthy Control Participants

In addition to those exclusion criteria already outlined above, control participants will also be excluded if they:

1. Have any current, or previous, diagnosis of any major psychiatric disorder, i.e. to include (but not limited to) mood, anxiety, and psychiatric disorders, or any substance-induced psychiatric disorders.
2. Have any first-degree relatives with history of psychosis likely related to schizophrenia, bipolar affective disorder, or schizoaffective disorder.
3. Have previously been diagnosed with a DSM-IV Axis II spectrum disorder.

Patient Participants

Patient patients will be excluded if they meet any of the criteria already outlined, and also if they:

1. Have experienced any changes in pharmacological treatment and dose in the 4 weeks preceding study enrollment.
2. We will exclude patients whose paranoid ideation might prevent them from feeling comfortable in the task- or scanning-environment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 159 (Actual)
Dates: Start 2005-03-08; Study Completion 2017-02-13

PRIMARY OUTCOMES:
Whether MRI responses in components of reward circuits are attenuated in patients, in the context of paradigms that require individuals to detect mismatches between expected & experienced outcomes, and to modify responses based on those... | one MRI

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Stein, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (2):
- United States (2):
  - University of Maryland, Baltimore, Baltimore, Maryland
  - National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland

REFERENCES:
- [Background] Addington D, Addington J, Schissel B. A depression rating scale for schizophrenics. Schizophr Res. 1990 Jul-Aug;3(4):247-51. doi: 10.1016/0920-9964(90)90005-r. PMID 2278986
- [Background] Akil M, Kolachana BS, Rothmond DA, Hyde TM, Weinberger DR, Kleinman JE. Catechol-O-methyltransferase genotype and dopamine regulation in the human brain. J Neurosci. 2003 Mar 15;23(6):2008-13. doi: 10.1523/JNEUROSCI.23-06-02008.2003. PMID 12657658
- [Background] Alain C, McNeely HE, He Y, Christensen BK, West R. Neurophysiological evidence of error-monitoring deficits in patients with schizophrenia. Cereb Cortex. 2002 Aug;12(8):840-6. doi: 10.1093/cercor/12.8.840. PMID 12122032